CLINICAL TRIAL: NCT02995395
Title: The Role of the Mucosal Impedance Balloon in the Diagnosis and Treatment Eosinophilic Esophagitis
Brief Title: Mucosal Impedance Balloon in Diagnosis and Treatment of Eosinophilic Esophagitis (EoE)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Sandhill Scientific (Industry)
Responsible Party: Principal Investigator, David A. Katzka, Principal Investigator, Mayo Clinic
Other Study IDs: 16-005863
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Eosinophilic Esophagitis; Healthy
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mucosal Impedance Balloon catheter: At the conclusion of the endoscopy, all fluids will be aspirated from the esophagus. The endoscope will then be left in place in the mid-esophagus and a custom Mucosal Impedance (MI) balloon assembly four axial arrays of 10 sensors (total of 40 sensors) will be positioned along the esophageal mucosal wall under direct visualization to directly measure MI at uniform intervals. Once in place, impedance readings will be recorded for a total of 2 minutes. At this point both the endoscope and impedance catheter will be withdrawn simultaneously.
  Interventions: Device: Mucosal Impedance Balloon catheter

INTERVENTIONS:
Device: Mucosal Impedance Balloon catheter — During the clinical endoscopy (a standard procedure that allows your doctor to look at the inside of your swallowing tube), the 2 mm catheter (tiny tube), called an Intraluminal Impedance Balloon, will be passed through the channel of the standard endoscope.
  o The catheter (tiny tube) will be placed through the endoscope in your esophagus (swallowing tube) for two minutes, readings from the catheter will be recorded.
  Other Names: Impedance balloon testing

SUMMARY:
This study will evaluate the role the balloon mucosal impedance may have in diagnosing and monitoring the patients with Eosinophilic Esophagitis. We will compare the results of the balloon mucosal impedance in patients with Eosinophilic esophagitis and controls.

DETAILED DESCRIPTION:
The standard diagnostic evaluation for EoE includes upper endoscopy with esophageal biopsies. Recently we completed the study "Mucosal impedance in eosinophilic esophagitis and the effect of treatment" using a new technology allowing for direct assessment of mucosal impedance at the time of routine upper endoscopy to assess esophageal integrity and disease activity and alevate the need for biopsies.

For this study, Sandhill Scientific has customized a Mucosal Impedance balloon (MI) assembly to provide precise measurements over a broad area of esophageal epithelium, while eliminating the fluids and spanning across a 10 mm luminal area using the same direct assessment as the mucosal impedance at the time of routine upper endoscopy.

ELIGIBILITY:
Inclusion criteria:

* Adults ages 18-90 undergoing clinically indicated upper endoscopy
* Patients with EoE, defined as dysphagia with histologic finding of greater than or equal to 15 eosinophils per high powered field on esophageal biopsy despite at least 6 weeks of twice daily proton pump inhibitor therapy
* Patients undergoing clinically indicated upper endoscopy for indications other than dysphagia or GERD with normal appearing esophageal mucosa.

Exclusion criteria:

* Medical conditions such as severe heart or lung disease that preclude safe performance of endoscopy
* Patients with conditions known to be associated with esophageal eosinophilia, including Crohn's disease, Churg-Strauss, achalasia, and hypereosinophilic syndrome
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Eosinophilic Esophagitis having an upper endoscopy. Patients having an upper endoscopy for dysphagia or GERD
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Diminished mucosal impedance in patients with Eosinophilic Esophagitis | 1 year
  Patient with eosinophilic esophagitis have diminished mucosal impedance, reflecting increased permeability to allergens occurring in the esophagus. The impedance measurements are also variable throughout the esophageal mucosa reflecting the patchy histology of eosinophilic esophagitis.

CONTACTS AND LOCATIONS:
Overall Officials: David A Katzka, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexander JA, Ravi K, Geno DM, Tholen CJ, Higginbotham TC, Wildhorn S, Camilleri M, Vaezi MF, Katzka DA. Comparison of mucosal impedance measurements throughout the esophagus and mucosal eosinophil counts in endoscopic biopsy specimens in eosinophilic esophagitis. Gastrointest Endosc. 2019 Apr;89(4):693-700.e1. doi: 10.1016/j.gie.2018.08.031. Epub 2018 Aug 24. PMID 30145316
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials